CLINICAL TRIAL: NCT05182034
Title: A Multi-center, Randomized, Double-Blinded, Active-Controlled, Phase II Clinical Trial to Evaluate Efficacy and Safety of SMUP-IA-01 in Patients With Knee Osteoarthritis
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of SMUP-IA-01 in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-SMUP-IA-01-P02
Record Dates: First submitted 2021-12-12; First posted 2022-01-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: human umbilical cord blood derived mesenchymal stem cells; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group 1: SMUP-IA-01 (low dose) (Experimental): Investigational Product - 4.0×10^6 cells/2 mL of SMUP-IA-01 (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(low dose)
- Study Group 2:SMUP-IA-01 (mid dose) (Experimental): Investigational Product - 1.0×10^7 cells/2 mL of SMUP-IA-01 (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(mid dose)
- Active Control Group (Active Comparator): Investigational Product - 2 ml of 1% sodium hyaluronate (2 ml of sodium chloride injection is administered before administration of 1% sodium hyaluronate)
  Interventions: Drug: Active Control Group Sodium chloride

INTERVENTIONS:
Biological: SMUP-IA-01(low dose) — A single knee administration of SMUP-IA-01(low-dose, 4.0 x 10^6 cells/2mL)
  Other Names: SMUP allogenic cord blood-derived mesenchymal stem cell (SMUP-Cell)
  Arms: Study Group 1: SMUP-IA-01 (low dose)
Biological: SMUP-IA-01(mid dose) — A single knee administration of SMUP-IA-01(mid-dose, 1.0 x 10^7 cells/2mL)
  Other Names: SMUP allogenic cord blood-derived mesenchymal stem cell (SMUP-Cell)
  Arms: Study Group 2:SMUP-IA-01 (mid dose)
Drug: Active Control Group Sodium chloride — A single knee administration of Sodium chloride
  Other Names: Sodium chloride
  Arms: Active Control Group

SUMMARY:
This clinical trial is for patients who have been diagnosed with Kellgren-Lawrence (K&L) Grade 2 or 3 knee osteoarthritis on radiographic examination. Only subjects who voluntarily agree to participate by filling out the written Informed Consent document will undergo screening for subject selection (inclusion/exclusion) criteria, at which time the severity of OA in each knee will be used to determined which knee will be treated (index knee - i.e., the more severely affected knee), and enroll in this study.

DETAILED DESCRIPTION:
Patients who meet the inclusion/exclusion criteria will be randomly assigned at visit 2 to either of study group 1(low-dose), study group 2 (mid-dose) or active control group at 1:1:1 ratio. Patients will be administered with investigational product. Investigational product will be administered into the to-be-treated (index) knee one time within 7 days after randomization.

All patients enrolled will be followed up a total of 6 times (1, 4, 8, 12, 24, and 52 weeks) for up to post-dose 12 months. The patients should visit the study facility according to the visit schedule, and will undergo safety evaluation (vital sign, laboratory test, etc.) and efficacy evaluation [Western Ontario and McMaster Universities osteoarthritis index (WOMAC), 100-mm visual analogue scale (VAS), International Knee Documentation Committee (IKDC) subjective knee evaluation].

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥ 19 years of age on the date on which the consent form was signed
2. Patients diagnosed with knee osteoarthritis in at least one knee according to the clinical and radiological definition criteria of American College of Rheumatology (ACR) guidline at screening visit
3. Patients with knee OA corresponding to K&L Grade 2 or 3 on radiographic examination at screening visit
4. Patients with less than 35 of BMI at screening visit
5. Patients who voluntarily decide to participate and sign the consent form
6. Patients who have persistent symptoms despite having undergone a reasonable trial of standard therapy (i.e., for a minimum of 3 months)

Exclusion Criteria:

1. Patients with any of the following diseases.

   - infectious arthritis, autoimmune or inflammatory joint diseases, gout, recurrent pseudogout, Paget's disease, intra-articular displaced fracture, ochronosis, acromegaly, haemochromatosis, Wilson's disease, genetic disease (hyperkinesia etc.), genetic collagen disorder, etc.
2. Patients who have ever undergone surgery or radiotherapy in the knee joint area within the 12 weeks prior to the screening visit date, or who have not been recovered from its side effect yet.
3. Patients with SIF (Subchondral insufficiency fracture) corresponding to type II of the RPOA (rapidly progressive osteoarthritis).
4. Patients whose physical examination results show severe degree of ligament instability.
5. Patients who have ever been given any intraarticular drug injection (i.e., hyaluronic acid injection, etc.) in to-be-treated (index) knee within the 6 months, prior to the screening visit date.
6. Patients who have ever been given steroids via intraarticular injection in to-be-treated (index) knee within the 12 weeks prior to the screening visit date.
7. Patients who have ever taken medications or given therapy below within the past 2 weeks on the basis of screening visit date. However, if patients have 14 days of wash-out period, the patient is allowed to participate.

   * drugs containing the ingredient of glucosamine, chondroitin sulfate, or diacerein
   * drugs containing herbal ingredient or herbal drugs for knee OA pain relief
   * anti-inflammatory analgesics or NSAIDs (prescription/non-prescription drugs). (However, patients who take acetaminophen and have 3 days of wash-out period are allowed to participate.)
   * oral steroids
   * hospital physiotherpy or oriental medicine treatment (buhang, acupunture, moxibustion etc.)
8. Patients who have skin disease on injection site or who are judged inappropriate for intra-articular injection on to-be-treated knee.
9. Patients who are judged unsuitable for MRI scanning (3.0 Tesla or higher) due to an insertion of metal material (i.e., heart pacemaker, cerebral aneurysm clip, etc.) or obstructive phobia. However, patients who have an insertion of metal material that is not affected by the magnetic field is allowed to participate
10. Patients with clinically significant past or present illness as follows;

    * heart diseases (i.e., myocardial infarction, coronary artery bypass surgery, arrhythmia and other serious heart diseases, etc.)
    * uncontrolled hypertension (not controlled down to 140/90 mmHg or below even after treatment with 3 or more antihypertensive drugs)
    * kidney disease (i.e., chronic kidney failure, glomerulonephritis, etc.)
    * liver disease (i.e., acute or chronic liver disease such as cirrhosis, fatty liver, etc.)
    * endocrine diseases (i.e., thyroiditis, diabetes insipidus, Cushing's disease, etc.)
    * other serious systemic diseases
11. Patient with ongoing autoimmune disorder that requires treatment with an immunosuppressive medication
12. Patients with infection that requires administration of parenteral antibiotics
13. Patients with a history of mental illness or epilepsy
14. Patients who have been diagnosed with cancer within the 5 years prior to the screening visit date
15. Patients who have been given immunosuppressive drugs such as cyclosporin A or azathioprine within the 6 weeks prior to the screening visit
16. Patients with a history of allergic reactions to hyaluronic acid injections, cryoprotectant (dimethyl sulfoxide, DMSO), or gentamicin.
17. Patients who are pregnant or lactating, or patients who have a plan to become pregnant during the study period
18. Male or female patients who do not agree to avoid pregnancy or the use of appropriate contraceptive methods during the study period. But women who have given infertility surgery or who have passed menopause one year or more are allowed to participate without the consent for contraception.
19. Patients who have been given any other cell therapy products or who plan to do so during the study period.
20. Patients who have been given any other investigational products including device within the 3 months prior to the screening visit date.
21. Patients who are judged by the investigator as inappropriate for enrollment into the study, for any reasons other than the reasons specified above.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Change in the WOMAC(Western Ontario and McMaster University Osteoarthritis Index) total score at post-dose 52 weeks from baseline | Baseline, 52 week
  Total score is between 0 point (no symptoms) ~ 96 points (higher score representing worse symptoms).

SECONDARY OUTCOMES:
Change amount of WOMAC total score at post-dose 24 weeks from the baseline | Baseline, 24 week
  Total score is between 0 point (no symptoms) ~ 96 points (higher score representing worse symptoms).
Chage amount of WOMAC score by item (pain, stiffness, physical function) at post-dose 24 weeks and 52 weeks from the baseline | Baseline, 24 week, 52 week
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68)
Chage amount of 100-mm VAS((Visual Analogue Scale) at post-dose 1 week, 4 weeks, 8 weeks, 12 weeks, 24 weeks and 52 weeks from the baseline | Baseline, 1 week, 4 week, 8 week, 12 week, 24 week, 52 week
  The score ranges from "0" or no pain to "100" very severe pain
Chage amount of IKDC(International Knee Documentation Committee) at post-dose 1 week, 4 weeks, 8 weeks, 12 weeks, 24 weeks and 52 weeks from the baseline | Baseline, 1 week, 4 week, 8 week, 12 week, 24 week, 52 week
  IKDC subjective knee evaluation consists of three categories:
  symptoms, sports activities, and functions. For each category, there are 7 questions for symptoms, 2 questions for sports activities, and 2 questions for functions, a total of 11 questions for evaluation. The scores for each category are summed up and divided into 87, which is the maximum score possible, and then is evaluated by converting it into a scale of 100 points. Higher score indicates better function and less symptoms for the knee.
Change in the WOMAS(whole-organ magnetic resonance imaging score) at post-dose 52 weeks from the baseline | Baseline, 52 week
  Total score is between 0 point (no symptoms) ~ 96 points (higher score representing worse symptoms).
Change in T2 mapping at post-dose 52 weeks from the baseline | Baseline, 52 week
  Changes on the knee structure through qualitative and quantitative evaluation of the collagen matrix of knee cartilage.
Change in K&L grade, joint space width, mechanical axis, and anatomical axis at post-dose 52 weeks from the baseline | Baseline, 52 week
  K & L grade (0 to 4 Grade): which means that the higher the grade, the greater the joint damage and the stenosis of the joint.
  Joint space width(mm): Evaluation of disease progression in target knee as ascertained by change from baseline joint space width (JSW) determined using radiography.
  Mechanical axis(Angle): A line connecting the femoral head center point and the ankle joint center point. Anatomical axis(Angle): The middiaphyseal line of the femur and tibia
Change amount of biomarkers at post-dose 1 week, 4 weeks, 8 weeks, 12 weeks, 24 weeks and 52 weeks against the baseline; serum CTX-I, Serum HA, Serum MMP-3, Urine CTX-I, Urine CTX-II. | baseline, 1 week, 4 week, 8 week, 12 week, 24 week, 52week
  serum C-terminal cross-linking telopetides of collagen type I(CTX-I), serum hyaluronan, serum matrix metalloproteinase-3 (MMP-3), urine C-terminal cross-linking telopetides of collagen type II (CTX -II), urine C-terminal cross-linking telopetides of collagen type I(CTX-I).
  Serum CTX-I, Serum HA, Serum MMP-3, Urine CTX-I, Urine CTX-II are reported in pg/ml.
Percentage of patients who took the rescue drugs and dosage at post-dose 1 week, 4 weeks, 8 weeks, 12 weeks, 24 weeks and 52 weeks | 1 week, 4 week, 8 week, 12 week, 24 week, 52week
  Subjects will receive Patient Diary, and use of the rescue drug should be recorded on the Patient Diary.

CONTACTS AND LOCATIONS:
Overall Officials: Myungchul Lee, MD, PhD, Principal Investigator — Seoul National University Hospital; Chonghyuk Choi, MD, PhD, Principal Investigator — Severance Hospital; Chongbum Chang, MD, PhD, Principal Investigator — Seoul Nation University Bundang Hospital; Seungbum Han, MD, PhD, Principal Investigator — Korea University Anam Hospital; Sunghwan Kim, MD, PhD, Principal Investigator — Gangnam Severance Hospital
Locations (5):
- South Korea (5):
  - Seoul Nation University Bundang Hospital, Gyeonggi-do
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospita, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul